CLINICAL TRIAL: NCT05224674
Title: Comparative Effects of Focused (Large Focused) and Radial (Controlled Unfocused) Shock-Wave Therapies in Hip Osteoarthritis.
Brief Title: Comparative Effects of Focused and Radial Shock-Wave Therapies in Hip Osteoarthritis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Volkan Şah, Principal Investigator, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Van Yuzuncu Yil University
Record Dates: First submitted 2022-01-18; First posted 2022-02-04 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Large-Focused Extracorporeal Shock Wave Therapy (Active Comparator)
  Interventions: Device: Extracorporeal Shock Wave Therapy (ESWT)
- Controlled-Unfocused Extracorporeal Shock Wave Therapy (Active Comparator)
  Interventions: Device: Extracorporeal Shock Wave Therapy (ESWT)
- Sham Extracorporeal Shock Wave Therapy (Sham Comparator)
  Interventions: Device: Extracorporeal Shock Wave Therapy (ESWT)

INTERVENTIONS:
Device: Extracorporeal Shock Wave Therapy (ESWT) — The ESWT device is product of Elettronica Pagani, Italy.

SUMMARY:
There is no scientific study in the literature regarding the use of shock wave therapy in hip osteoarthritis. In this study, we aim to investigate both the effectiveness of ESWT and which type of ESWT can be more effective in hip osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* unilateral or bilateral hip osteoarthritis

Exclusion Criteria:

* other disorders that are contraindications for shockwave therapy, not have received ESWT treatment before

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | at baseline.
  patient's self-assessment of pain, in the range of 0 to 10, higher scores mean a worse outcome.
Visual Analogue Scale (VAS) | 4 weeks after baseline.
  patient's self-assessment of pain, in the range of 0 to 10, higher scores mean a worse outcome
Visual Analogue Scale (VAS) | 8 weeks after baseline.
  patient's self-assessment of pain, in the range of 0 to 10, higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | at baseline.
  24-item questionnaire for osteoarthritis, in the range of 0 to 96, higher scores mean a worse outcome
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 4 weeks after baseline.
  24-item questionnaire for osteoarthritis, in the range of 0 to 96, higher scores mean a worse outcome
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 8 weeks after baseline.
  24-item questionnaire for osteoarthritis, in the range of 0 to 96, higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Volkan Şah, Principal Investigator — Yüzüncü Yıl Üniversitesi Tıp Fakültesi
Locations (1):
- Volkan Şah, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No